CLINICAL TRIAL: NCT02519946
Title: On-Line Intervention to Lower Cardiovascular Risk in Pediatric Heart Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Seda Tierney, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15GRNT25680030
Record Dates: First submitted 2015-07-30; First posted 2015-08-11 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Vascular; Change; Dietary Modification; Physical Activity; Health Behavior; Attitude to Health
Keywords: Heart Transplantation; Tonometry; Exercise Test; Diet; Cardiovascular Physiology; Telemedicine; Pediatrics; Health Behavior; Physical Fitness; Exercise Movement Techniques; Adolescent Behavior; Child Behavior
MeSH Terms: conditions — Motor Activity; Health Behavior; Adolescent Behavior; Child Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- On-Line Diet and Exercise Intervention (Experimental)
  Interventions: Other: On-Line Diet and Exercise Intervention

INTERVENTIONS:
Other: On-Line Diet and Exercise Intervention — Initial 16 weeks of on-line, live exercise instruction 3x/week and on-line, diet sessions followed by 16 weeks of weekly exercise and diet sessions.

SUMMARY:
Pediatric heart transplant patients have a high-risk cardiovascular profile affecting their long-term outcomes and survival. Currently, no effective cardiovascular preventative care is provided for this pediatric population, in part, due to the fact that clinic-based programs are not easily accessible to children and their families. However, tele-health has been show to improve medical outcomes by making care more accessible to these patients. This study aims to meet the urgent need for an effective and sustainable delivery of preventative care to pediatric heart transplant patients using a diet and exercise intervention program delivered live over the internet direct to these patients' homes.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant >11 months before baseline visit
* Able to fast overnight
* Cardiac clearance to exercise by the primary cardiologist
* Presence of an adult at home during the exercise training sessions for patients < 14 years of age

Exclusion Criteria:

* Acute illness
* Latex allergy
* Document transplant rejection < 3 months
* Re-transplantation or multi-organ transplantation
* Malignancy

Ages: 9 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2015-08; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Endothelial Pulse Amplitude Testing Index | Baseline, 16 weeks, and 32 weeks
  Test of endothelial function

SECONDARY OUTCOMES:
Arterial Tonometry | Baseline, 16 weeks, and 32 weeks
Carotid Artery Imaging | Baseline, 16 weeks, and 32 weeks
Fasting Low-Density Lipoprotein Level | Baseline, 16 weeks, and 32 weeks
Volume of Oxygen Consumed at Maximal Exertion | Baseline, 16 weeks, and 32 weeks
Physical and Psychosocial Health Questionnaire Scores | Baseline, 16 weeks, and 32 weeks
  Both parents and patients will be asked to complete this questionnaire
Functional Movement Screening Score | Baseline, 16 weeks, and 32 weeks
  Participants will be asked to perform certain movements. The range of motion will be scored and totaled for evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Seda Selamet Tierney, MD, Principal Investigator — Stanford Children's Hospital
Locations (1):
- Stanford Children's Health, Palo Alto, California, United States

REFERENCES:
- [Derived] Chen AC, Ramirez FD, Rosenthal DN, Couch SC, Berry S, Stauffer KJ, Brabender J, McDonald N, Lee D, Barkoff L, Nourse SE, Kazmucha J, Wang CJ, Olson I, Selamet Tierney ES. Healthy Hearts via Live Videoconferencing: An Exercise and Diet Intervention in Pediatric Heart Transplant Recipients. J Am Heart Assoc. 2020 Feb 4;9(3):e013816. doi: 10.1161/JAHA.119.013816. Epub 2020 Jan 24. PMID 31973598